CLINICAL TRIAL: NCT01870700
Title: The Effect of Lactobacillus Reuteri Supplementation to Adult With Functional Chronic Constipation: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Lactobacillus Reuteri in Adult With Functional Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catholic University, Italy (Other)
Responsible Party: Principal Investigator, veronica ojetti, adjunt professor, Catholic University, Italy
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: no one
Record Dates: First submitted 2013-05-25; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Functional Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lactobacillus reuteri (Experimental): Intervention: supplementation with the probiotic Lactobacillus reuteri (DSM 17938),Reuflor, was administered in the dose of 108 colony-forming units (CFU) in tablets of a commercially available preparation (Reuflor, Italchimici, Pomezia; BioGaia AB, Stockholm, Sweden), 30 minutes after feeding, twice per day for 4 weeks.
  Interventions: Drug: lactobacillus reuteri
- placebo (Placebo Comparator): a supplementation with placebo was administered in tablets of a commercially available preparation 30 minutes after feeding, twice per day for 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lactobacillus reuteri — Lactobacillus reuteri (DSM 17938) was administered in the dose of 108 colony-forming units (CFU) in tablets of a commercially available preparation (Reuflor, Italchimici, Pomezia; BioGaia AB, Stockholm, Sweden), 30 minutes after feeding, twice per day for 4 weeks
  Other Names: Reuflor
  Arms: lactobacillus reuteri
Drug: placebo — a supplementation with placebo was administered in tablets of a commercially available preparation 30 minutes after feeding, twice per day for 4 weeks
  Arms: placebo

SUMMARY:
A double-blind, placebo Randomized Controlled Trial, To evaluate the effects of L. reuteri in adult patients with functional constipation.

DETAILED DESCRIPTION:
Patients affected by functional constipation according to Rome III criteria. The increase of Bowel Movements/week frequency was the primary outcome, while the improvement of stool consistency was the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* functional constipation rome III

Exclusion Criteria:

* hypothyroidism or other metabolic or renal abnormalities, or
* antibiotic's treatment,
* probiotic or prebiotic supplementation in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The increase of BMs/week frequency | January to June 2012 (up to 6 months)

SECONDARY OUTCOMES:
the improvement of stool consistency | january to june 2012 (up to 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: veronica ojetti, Study Chair — catholic university
Locations (1):
- Catholic University Sacred Heart, Rome, Italy/rome, Italy

REFERENCES:
- [Background] Coccorullo P, Strisciuglio C, Martinelli M, Miele E, Greco L, Staiano A. Lactobacillus reuteri (DSM 17938) in infants with functional chronic constipation: a double-blind, randomized, placebo-controlled study. J Pediatr. 2010 Oct;157(4):598-602. doi: 10.1016/j.jpeds.2010.04.066. Epub 2010 Jun 12. PMID 20542295
- [Derived] Ojetti V, Ianiro G, Tortora A, D'Angelo G, Di Rienzo TA, Bibbo S, Migneco A, Gasbarrini A. The effect of Lactobacillus reuteri supplementation in adults with chronic functional constipation: a randomized, double-blind, placebo-controlled trial. J Gastrointestin Liver Dis. 2014 Dec;23(4):387-91. doi: 10.15403/jgld.2014.1121.234.elr. PMID 25531996